CLINICAL TRIAL: NCT01381822
Title: A Phase 1 Dose-Escalation Study to Determine the Safety of TH-302 in Combination With Sunitinib in Patients With Advanced Renal Cell Carcinoma,Gastrointestinal Stromal Tumors and Pancreatic Neuroendocrine Tumors
Brief Title: Dose-Escalation Study of TH-302 in Combination With Sunitinib to Treat Patients With Advanced Renal Cell Carcinoma,Gastrointestinal Stromal Tumors and Pancreatic Neuroendocrine Tumors
Acronym: TH-CR-410
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Threshold Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-CR-410
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Advanced Renal Cell Carcinoma; Gastrointestinal Stromal Tumors; Pancreatic Neuroendocrine Tumors
Keywords: TH-302; Advanced Renal Cell Carcinoma; RCC; Gastrointestinal Stromal Tumors; GIST; Phase 1; Sunitinib; Pancreatic Neuroendocrine Tumors; PNET
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Neuroectodermal Tumors, Primitive | interventions — TH 302

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TH-302 Dose escalation (Experimental): The initial dose of TH-302 will be 240 mg/m2. A Dose Level minus 1 and 2 will be built into the study in the event that subjects experience excessive toxicity at Dose Level 1. Dose escalation will continue with approximately 40% increases from the previous dose level; however lower dose increases of 20-39% may be implemented after consultation between the Investigators, Medical Monitor and Sponsor with the percent increase dependent on the current dose level and the cumulative safety data.
  Interventions: Drug: TH-302

INTERVENTIONS:
Drug: TH-302 — TH-302: administered by IV infusion over 30 or 60 minutes on Days 8, 15 and 22 of a 42 day cycle.

SUMMARY:
The primary objectives are:

Dose escalation:

1. To determine the MTD and DLT(s) of TH-302 when used in combination with sunitinib.

Dose expansion:

1. To make a preliminary assessment of the efficacy of TH-302 in combination with sunitinib as determined by the response rate and the progression-free survival in subjects with advanced RCC treated at the RP2D
2. To assess the safety of TH-302 in combination with sunitinib and determine a recommended Phase 2 dose of the combination.

The secondary objectives are:

Dose expansion:

1. To make a preliminary assessment of the efficacy of TH-302 in combination with sunitinib as determined by stable disease or better rate, duration of response and overall survival in subjects with advanced RCC treated at the RP2D.

The exploratory objective is:

1. To explore the association of serum hypoxia biomarkers with efficacy endpoints.

DETAILED DESCRIPTION:
This Phase 1 dose-escalation study will use a classic dose escalation design to determine the MTD of TH-302 when used in combination with sunitinib. The study will be divided into two parts completed in succession to determine the recommended phase 2 dose (RP2D) for dose expansion.

Part A:

The dose of TH-302 will be escalated in cohorts of 3-6 subjects. The initial dose of TH-302 will be 240 mg/m2. A Dose Level minus 1 and 2 will be built into the study in the event that subjects experience excessive toxicity at Dose Level 1. Dose escalation will continue with approximately 40% increases from the previous dose level; however lower dose increases of 20-39% may be implemented after consultation between the Investigators, Medical Monitor and Sponsor with the percent increase dependent on the current dose level and the cumulative safety data.

If a subject experiences a DLT, 3 additional subjects will be enrolled at that dose level for a total of 6 subjects in that cohort. If no additional DLTs are observed, dose escalation will resume. However, if 2 or more of 6 subjects within a cohort experience a DLT, that dose will be considered to exceed the MTD. The MTD will then be defined at the next lower dose level whereby 6 subjects were treated and < 1 subject experienced a DLT. The maximum dose of TH-302 will be 575 mg/m2.

The MTD will be based on toxicities occurring during the first cycle.

TH-302 will be administered by IV infusion over 30-60 minutes on Days 8, 15 and 22 of a 42-day cycle (6 weeks).

The dose of sunitinib will remain fixed: 50 mg administered PO daily on days 1 to 28 day of a 42-day cycle (6 weeks). On days when both sunitinib and TH-302 are administered, sunitinib should be administered at least 2 hours before or at least 2 hours after completion of the TH-302 dose.

Part B:

Once the MTD from Part A has been determined, Part B can commence.

The initial dose of TH-302 will be one dose level higher than the MTD established in Part A. The dose of TH-302 will be escalated in cohorts of 3-6 subjects. A Dose Level at the MTD established in Part A will be built into the study in the event that subjects experience excessive toxicity at the initial dose. Dose escalation will continue with approximately 40% increases from the previous dose level; however lower dose increases of 20-39% may be implemented after consultation between the Investigators, Medical Monitor and Sponsor with the percent increase dependent on the current dose level and the cumulative safety data.

If a subject experiences a DLT, 3 additional subjects will be enrolled at that dose level for a total of 6 subjects in that cohort. If no additional DLTs are observed, dose escalation will resume. However, if 2 or more of 6 subjects within a cohort experience a DLT, that dose will be considered to exceed the MTD. The MTD will then be defined at the next lower dose level whereby 6 subjects were treated and < 1 subject experienced a DLT.

The MTD will be based on toxicities occurring during the first cycle.

TH-302 will be administered by IV infusion over 30-60 minutes on Days 8, 15 and 22 of a 42-day cycle (6 weeks).

The dose of sunitinib will remain fixed: 37.5 mg administered PO daily on days 1 to 28 of a 42-day cycle (6 weeks).

On days when both sunitinib and TH-302 are administered, sunitinib should be administered at least 2 hours before or at least 2 hours after completion of the TH-302 dose.

An additional 10 RCC subjects will be enrolled at the recommended phase 2 dose (RP2D) for the dose expansion portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's IRB/Ethics Committee
* Pathologically confirmed diagnosis of

  * advanced RCC or
  * GIST after disease progression on or intolerance to imatinib mesylate (dose escalation only)
  * Unresectable locally advanced or metastatic pancreatic neuroendocrine tumors (dose escalation only)
* Recovered from reversible toxicities of prior therapy
* Evaluable disease by RECIST criteria (at least one target or non-target lesion for dose escalation cohorts; at least 1 target lesion for dose expansion cohort)
* ECOG performance status of 0 - 2
* Life expectancy of at least 3 months
* Acceptable liver function:

  * Bilirubin less than or equal to 1.5 times upper limit of normal (ULN)
  * AST (SGOT) and ALT (SGPT) less than or equal to 3.0 times ULN
* Acceptable renal function:

  * Serum creatinine ≤ Upper Limit Normal,
* Acceptable hematologic status (without hematologic support):

  * ANC greater than or equal to 1500 cells/μL
  * Platelet count greater than or equal to 100,000/μL
  * Hemoglobin great than or equal to 9.0 g/dL
* Acceptable cardiac function:

  * Normal 12-lead ECG (clinically insignificant abnormalities permitted)
  * LVEF normal by MUGA or echocardiogram
* Urinalysis: No clinically significant abnormalities
* Acceptable thyroid function
* All women of childbearing potential must have a negative serum pregnancy test and all subjects must agree to use effective means of contraception (surgical sterilization or the use or barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 6 months after the last dose

Exclusion Criteria:

* Prior therapy with more than 2 myelosuppressive cytotoxic chemotherapy regimens (does not include neoadjuvant and adjuvant therapy)
* Current use of drugs with known cardiotoxicity or known interactions with sunitinib (see product label)
* Anticancer treatment with radiation therapy, chemotherapy, targeted therapies (erlotinib, lapatinib, etc.), immunotherapy, hormones or other antitumor therapies within 3 weeks prior to study entry (6 weeks for nitrosoureas or mitomycin C)
* Significant cardiac dysfunction:

  * Cardiac events within 12 months prior to treatment including MI and severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic CHF, cerebrovascular accident or transient ischemic attack or pulmonary embolism
  * > Grade 2 QTc prolongation
  * Requirement for antiarrhythmics
  * Uncontrolled arrhythmias within the past 6 months
  * Angina pectoris requiring antianginal medication within the past 6 months
  * Clinically significant valvular heart disease
  * Poorly controlled hypertension despite adequate blood pressure medication
* Seizure disorders requiring anticonvulsant therapy
* Known brain metastases (unless previously treated and well controlled for a period of greater than or equal to 3 months)
* Other active malignancy, except for adequately treated non-melanoma skin cancer, in situ cancer
* Severe chronic obstructive or other pulmonary disease with hypoxemia (requires supplementary oxygen, symptoms due to hypoxemia or oxygen saturation <90% by pulse oximetry after a 2 minute walk) or in the opinion of the investigator any physiological state likely to cause normal tissue hypoxia
* Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1, without complete recovery
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Prior therapy with an hypoxic cytotoxin
* Subjects who participated in an investigational drug or device study within 21 days prior to study entry
* Known infection with HIV or active infection with hepatitis B or hepatitis C
* Subjects who have exhibited allergic reactions to a structural compound or biological agent similar to TH-302
* Females who are pregnant or breast-feeding
* Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
* Unwillingness or inability to comply with the study protocol for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
To determine the MTD and DLT(s) of TH-302 when used in combination with sunitinib. | Two years

SECONDARY OUTCOMES:
To make a preliminary assessment of the efficacy of TH-302 in combination with sunitinib as determined by the response rate and the progression-free survival in subjects with advanced RCC treated at the RP2D. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Starodub, MD, Principal Investigator — IU Health Goshen Center for Cancer Care; Mohammed Milhem, MD, Principal Investigator — University of Iowa
Locations (2):
- United States (2):
  - IU Health Goshen Center for Cancer Care, Goshen, Indiana
  - University of Iowa, Iowa City, Iowa

REFERENCES:
- See also: Threshold Pharmaceuticals Company Website — http://www.thresholdpharm.com/